

### RESEARCH SUBJECT INFORMATION CONSENT and AUTHORIZATION FORM

TITLE OF PROJECT:

Video and Temporal Spatial Parameters Assessment of Gait

after Dysport Treatment: A Pilot Study

NAME OF PRINCIPAL INVESTIGATOR:

Alberto Esquenazi, MD

AFTER HOURS PHONE:

PRINCIPAL INVESTIGATOR'S PHONE:

(215) 663-6667

(215) 663-6000

Support/Funding Statement:

pharmaceutical company. Funding to support the conduct of this study is being provided by Ipsen Biopharmaceuticals Inc., а

## WHAT IS A CONSENT FORM?

informed consent and includes: this study. This process of learning and thinking about a study before you make a decision is known as decision about whether to participate, you should understand the possible risks and benefits related to You are being asked to take part in a medical research study. Before you can make a knowledgeable

- Receiving detailed information about this research study;
- questions, you should ask for an explanation before you sign this form; decided to participate. If you don't understand something about the study or if you have Being asked to read, sign, and date this consent form, once you understand the study and have
- Being given a copy of your signed and dated consent form to keep for your own records

experimental drug, device, or procedure being studied and with the understanding that you may or may not benefit from your participation in the study. You should ask questions of the study doctor if you want The study doctor treats all subjects according to a research plan to obtain information about the family doctor. Your family doctor treats your specific health problem with the goal of making you better. to know more about this The relationship that you have with the study doctor is different than the relationship you have with your

## PURPOSE OF THE STUDY:

observation in lower limb spasticity as another technique to guide clinicians in identifying targeted muscles but they are not always available or effective. The purpose of this study is to evaluate the usefulness of video There are techniques available to identify targeted muscles for spasticity treatment with medication injection, for spasticity treatment with medication injection.

and your treating physician identified you as a candidate to receive spasticity medication injections You are being asked to participate in this study because you have ankle/foot spasticity; may use a leg brace

We plan to have up to 15 patients enrolled at MossRehab

60 Township Line Road

Elkins Park, PA 19027

Einstein.edu

Willowcrest

Einstein Medical Center Montgomery 1 of 6

# **DESCRIPTION OF PROCEDURES:**

scheduled 4-6 weeks after the first visit. Each visit will last about an hour. To take part, you must agree Taking part in this study will involve two to three visits to the clinic. The follow-up final visit will be

- Allow collection of information from you and your medical record about your medical history;
- Agree to be videotaped when you walk on at mat;
- If you do not want to be videotaped, you will not be able to take part in this study
- Agree to receive a spasticity treatment injection medication called Dysport
- muscles, causing a temporary reduction in muscle activity spasticity in adult patients. It is a botulinum toxin that blocks nerve activity in the treatment of spasticity. Dysport for injection is indicated for the treatment of lower limb Dysport is a medication currently used in clinical care that is FDA approved for the

## Screening/Baseline Visit

A member of the study will:

- Review demographics (gender, date of birth/age, ethnicity, race, height and weight)
- Review your medical/surgical history, including ongoing medical history
- Review your spasticity injection treatment history
- Review your current medications and allergies
- moving your ankle quickly from toe pointing down to toe pointing up and documenting the Measure your ankle and knee passive range of motion (PROM), tone with the Modified Ashworth Scale (MAS) and spasticity with the Tardieu Scale (TS). This entails the examiner
- comfortable walking speed and at your fast walking speed Ask you to walk and be videotaped walking with and without your shoes at your most

which muscles will be injected with the study medication Dysport. After the above is completed, the study doctor will review the videotape of you walking and decide

- The study doctor will inject the study medication in the targeted location(s) in your ankle/foot
- You will receive a minimum of 1000 units, but no more than 1500 units of the study medication.

team immediately. weeks. Should you have any problems related to the study visit or the injection, you may call the study Once the study medication is injected, an appointment for your follow-up visit will be made in 4-6

determines that is appropriate You may need to return for a second visit to complete the baseline procedures if the study doctor

### Follow-up Final Visit

A member of the study team will:

- feel walking, how your brace feels; how your foot feels. Talk to you about your experience after your injection such as how you feel generally; how you
- Review your medications

- Measure your ankle and knee PROM, MAS and TS
- Record video of your walking with and without shoes at your most comfortable walking speed and fast walking speed (MV) for observation and review

### Withdrawal Visit

If for some reason, your participation ends before you return for the follow-up visit, we will contact you to collect the following information to include with your research record:

Your general health; how you feel walking, how your brace feels; how your foot feels

### RISKS/DISCOMFORTS

Once you receive the injection, you may experience tenderness, soreness and bruising at the injection site.

nasopharyngitis (runny nose or sore throat), joint or muscle pain, dizziness and falls. After the injection, you may experience temporary adverse reactions such as: muscle weakness,

walkway mat has parallel bars to minimize this from occurring. During video observation of your walking, there is a risk of loss of balance, tripping, and/or falling. The

or Norplant. Also, you should not participate in this study if you are nursing an infant. partner should be using oral contraceptives, a barrier method of contraception, an intrauterine device (IUD), The risks to an unborn child or fetus are not known at this time. If you are sexually active, you and your

# **COSTS FOR STUDY PROCEDURES:**

participating in the study, you will receive the study medication Dysport at no cost to you. The cost for your routine medical care will be your or your insurance's responsibility. While you are

medical care for spasticity treatment. However, the cost of Dysport will be your or your insurance's Once your participation in the study has ended, you can still receive treatment with Dysport as part of your responsibility.

#### BENEFITS:

knowledge we gain may aid clinicians in improving treatment choices and outcomes for patients in There may be no personal benefit to you, but the knowledge received may be of value to humanity. The

### **ALTERNATIVES:**

targeted injection sites such as electrical stimulation, ultrasound and EMG. Alternative procedures or treatments for your condition are to continue with current standard of care, which may include Dysport or other botulinum toxins such as Botox and using other methods to aid in identifying

#### RIGHTS:

take part, you can change your mind at any time and stop taking part in the study. Whatever decision you make, it will not affect your care or the relationship you have with your doctors or the Albert Einstein Your participation is voluntary. You can choose to take part or not to take part in the study. If you choose to Healthcare Network.

You will be told of any new information learned during the course of the study which might affect your

understanding of the information in this consent and your willingness to continue to participate

Your participation in this study may be ended by the principal investigator or the sponsor if they feel it is in

No guarantees have been made as to the results of your participation in the study

# **COMPENSATION FOR INJURY:**

appropriate medical care for that injury within the capabilities of the Network. However, Albert Einstein the costs incurred may, ultimately, be your responsibility. Healthcare Network cannot assure that the medical care and treatment will be provided without charge, and In the event of an injury resulting from your participation in this project, you will be provided with clinically

# **CONFIDENTIALITY / AUTHORIZATION:**

summary of the results. You can search this Web site at any time Law. This Web site will not include information that can identify you. At most, the Web site will include a description of this clinical trial will be available on http://www.ClinicalTrials.gov as required by U.S.

use health information about you that we create, collect, or use as part of the research. This permission is called an Authorization. The federal Health Insurance Portability and Accountability Act (HIPAA) requires us to get your permission to

By signing this form, you authorize the use and sharing of the following information for this research:

- Information from your medical records that is necessary for this study (initials, date of birth, age weight, height and race)
- Information we collect from you about your medical history
- Clinical and research observations made during your participation in the research

study doctor. Your personal information will be removed and will be replaced by a unique number (coded) assigned by your

for drug and alcohol abuse unless specified above information related to genetic testing, treatment for AIDS/HIV, psychiatric care and treatment, or treatment Any health information that is used or shared under this Authorization will  ${\tt NOT}$  include any special health

(Ipsen Biopharmaceuticals Inc.). information for purposes related to this research: members of the research team and the funding source By signing this form, you authorize the following persons and organizations to receive your protected health

Healthcare Network and its Institutional Review Board (IRB), which is the committee responsible for ensuring they feel it necessary, identify you as a subject. your welfare and rights as a research participant, may review and/or photocopy study records which may, if (FDA) or the Office of Human Research Protections (OHRP) or the appropriate offices of Albert Einstein In addition, regulatory agencies that provide research oversight such as the Food and Drug Administration

If information obtained in the study is published, it will not be identifiable as your results unless you give specific permission.

4 of 6

and Accountability Act of 1996 and its privacy regulations and all other applicable laws that protect your information. A copy of the Notice will be provided to you. Notice of Privacy Practices (a separate document) provides more information on how we protect your possibility that your information could be used or disclosed in a way that it will no longer be protected. Our privacy. We will protect your information according to these laws. The Albert Einstein Healthcare Network complies with the requirements of the Health Insurance Portability Despite these protections, there

the study investigator at: for this study will not expire unless you cancel it. You can cancel this Authorization at any time by writing to The information collected during your participation in this study will be kept indefinitely. Your Authorization

Alberto Esquenazi, MD MossRehab 60 Township Line Rd. Elkins Park, PA 19027

cancelled the Authorization. However, no new information will be collected about you after you cancel the investigator and the research team may continue to use information about you that was collected before you If you cancel your Authorization, you will not be able to continue to participate in this research. The principal Authorization

but refusing to sign will not affect your health care outside the study. You have a right to refuse to sign this form. If you do not sign the form, you may not be in the research study,

## WITHDRAWAL FROM STUDY:

records follow-up, and all clinical data, as it relates to the study, will continue to be collected from your medical In the event that you withdraw from the study, the study physician will ask your permission to continue study

## **CONTACT INFORMATION:**

(215) 456-3517 or privacy@einstein.edu. you can contact the Network's Privacy Office at: Gratz Building, 1000 West Tabor Rd, Philadelphia, PA 19141, health information or if you feel the privacy of your health information has not been adequately protected, If you feel that you have not been adequately informed of your rights with respect to the privacy of your

that injury will be answered by Alberto Esquenazi, MD or his/her designate who can be reached at (215) 663-All questions regarding your participation in this study, or in the event of injury, all questions pertaining to

of the Institutional Review Board, Albert Einstein Healthcare Network, Paley Bldg., First Floor, (215) 456-6243 For any questions pertaining to your rights as a research subject, you may contact Robert Wimmer, MD, chair

# **UNDERSTANDING OF PARTICIPATION:**

time. Whenever I ask questions, the questions will be answered by a qualified member of the research been answered. I have been encouraged to ask questions about any aspect of this research study at any staff or by the investigator(s) listed on the first page of this consent form The information in this consent form has been explained to me and all of my current questions have

be given to me. By signing this form, I agree to participate in this research study and give authorization to use the information collected for this research as explained in this consent form. A copy of this consent form will

| Printed Name of Subject |
|---|
| Subject Signature (relationship, if kin or guardian signs for subject) Date: |
| Printed Name of Person Holding Consent Discussion |
| Signature of Person Holding Consent Discussion Date: |
| Witness to consent when applicable: |
| Witness Statement: Your signature indicates that you were present during the informed consent discussion of this research for the above named participant, that the information in the consent form and any other written information was verbally discussed with the participant (or legally authorized representative) in a language that he/she could understand, that he/she was given the chance to ask and receive answers to his/her questions, that the decision to take part in the research was freely made by the participant (or legally authorized representative) who indicated his/her consent and authorization to take part in this research by: |
| <ul><li>Signing his/her name</li><li>By making his/her mark</li><li>Other means:</li></ul> |
| of |
| WITNESS SIGNATURE:TIME:TIME: |
| INVESTIGATOR'S STATEMENT I, the undersigned, certify that to the best of my knowledge, the subject signing this consent form has had the study fully and carefully explained by me or a member of the study staff and has been given an opportunity to ask any questions regarding the nature, risks, and benefits of participation in this research study. |
| INVESTIGATOR OR DESIGNEE*: Date: |
| SIGNATURE |

Einstein Date: 26 Mar 2019

Albert Einstein Healthcare Network

\*DESIGNEE REFERS TO CO-INVESTIGATOR OR SUB-INVESTIGATOR ONLY.